CLINICAL TRIAL: NCT03386474
Title: A 24-week, Double-masked, Multicenter, Two-arm Extension Study to Collect Safety and Efficacy Data on Brolucizumab 6 mg Drug Product Intended for Commercialization in Patients With Neovascular Age-related Macular Degeneration Who Have Completed the CRTH258A2301 Study
Brief Title: Study of Safety and Efficacy of Brolucizumab 6 mg Drug Product Intended for Commercialization in Patients With nAMD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRTH258A2301E1
Record Dates: First submitted 2017-12-11; First posted 2017-12-29 (Actual); Results first posted 2020-04-30 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-03

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: double-masked, extension study; neovascular age-related macular degeneration; intravitreal injection; brolucizumab; aflibercept
MeSH Terms: interventions — brolucizumab; aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brolucizumab (Experimental): Brolucizumab 6 mg solution for IVT injection, single injection at Day 1 (baseline), Week 8, and Week 16 or Week 20
  Interventions: Drug: Brolucizumab 6 mg
- Aflibercept (Other): Aflibercept 2 mg solution for IVT injection, single injection at Day 1 (baseline), Week 8 and Week 16 to maintain the masking of the extension trial only.
  Interventions: Drug: Aflibercept 2 mg

INTERVENTIONS:
Drug: Brolucizumab 6 mg — Administered as opthalmic solution for an intravitreal injection to the study eye
  Other Names: RTH258
  Arms: Brolucizumab
Drug: Aflibercept 2 mg — Administered as an opthalmic solution for intravitreal injection to the study eye
  Other Names: EYELEA
  Arms: Aflibercept

SUMMARY:
The purpose of this extension study was to assess the safety and efficacy of the new formulation of brolucizumab 6 mg ophthalmic solution when given to the same patients who received brolucizumab in the core trial CRTH258A2301 (also known as CRTH258-C002). The medical condition treated in the core and extension trials was neo-vascular age-related macular degeneration (nAMD).

DETAILED DESCRIPTION:
Subjects in the United States who had completed the 96 week core trial, CRTH258A2301 (also referred as CRTH258-C002), were eligible to participate in the extension trial provided the core trial Visit 26 at week 96, was less than or equal to 12 weeks from the Baseline Visit in the extension trial, CRTH258A2301E1.

Subjects who were treated with aflibercept during the core trial and met the eligibility requirements of this extension trial continued to receive aflibercept in this extension trial in order to maintain the masking during the extension trial. No hypothesis testing or descriptive analyses were planned.

Subjects who were treated in the core trial with brolucizumab 3mg or brolucizumab 6 mg, and met the eligibility requirements of this extension trial, received the new formulation of brolucizumab 6 mg solution in the extension trial.

Enrolled subjects were to receive three intravitreal (IVT) ophthalmic injections. The study eye was the same eye that received the treatment in the core study. The extension trial consisted of 7 study visits at 4 week intervals over a period of 24 weeks.

Assessment of the efficacy and safety of brolucizumab 6 mg was based on a within-patient comparison with the last 6 months of corresponding core-study efficacy and safety data serving as the reference. Neither the patient selection process nor expected sample sizes supported a valid comparison between aflibercept and brolucizumab. The aflibercept arm was included only to maintain the masking in the extension trial. Data was presented descriptively for only brolucizumab in line with the study objective. No formal hypothesis testing was planned.

ELIGIBILITY:
Inclusion Criteria:

* Sign written informed consent
* Completed the core study, CRTH258A2301, also known as CRTH258-C002 as defined by assessments at Visit 26/Week 96 within ≤12 weeks of the baseline.

Exclusion Criteria:

* Patient discontinued the treatment or the core study prematurely at any time
* Patient received standard of care treatment for nAMD after completion of the core study
* Pregnant or nursing women and women of child-bearing potential
* Stroke or MI (myocardial infarction) within 3 months of the baseline extension visit

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-09-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (61):
- United States (59):
  - Novartis Investigative Site, Peoria, Arizona
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Arcadia, California
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, La Jolla, California
  - Novartis Investigative Site, Loma Linda, California
  - Novartis Investigative Site, Mountain View, California
  - Novartis Investigative Site, Oakland, California
  - Novartis Investigative Site, Redlands, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Golden, Colorado
  - Novartis Investigative Site, Bridgeport, Connecticut
  - Novartis Investigative Site, New London, Connecticut
  - Novartis Investigative Site, Altamonte Springs, Florida
  - Novartis Investigative Site, Deerfield Beach, Florida
  - Novartis Investigative Site, Fort Myers, Florida
  - Novartis Investigative Site, Ocala, Florida
  - Novartis Investigative Site, Palm Beach Gardens, Florida
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Tallahassee, Florida
  - Novartis Investigative Site, Vero Beach, Florida
  - Novartis Investigative Site, Winter Haven, Florida
  - Novartis Investigative Site, Boise, Idaho
  - Novartis Investigative Site, Bloomington, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Leawood, Kansas
  - Novartis Investigative Site, Shawnee Mission, Kansas
  - Novartis Investigative Site, Portland, Maine
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Waldorf, Maryland
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Reno, Nevada
  - Novartis Investigative Site, Toms River, New Jersey
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Shirley, New York
  - Novartis Investigative Site, Syracuse, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Southern Pines, North Carolina
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Dublin, Ohio
  - Novartis Investigative Site, Fairfield, Ohio
  - Novartis Investigative Site, Camp Hill, Pennsylvania
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Abilene, Texas
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Plano, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Warrenton, Virginia
  - Novartis Investigative Site, Silverdale, Washington
  - Novartis Investigative Site, Spokane, Washington
  - Novartis Investigative Site, University Place, Washington
  - Novartis Investigative Site, Morgantown, West Virginia
  - Novartis Investigative Site, Milwaukee, Wisconsin
- Puerto Rico (2):
  - Novartis Investigative Site, Arecibo
  - Novartis Investigative Site, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=293

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 150 subjects who completed the 96 week CORE trial (RTH258-C001) were eligible to continue in the extension. 62 CORE sub. were treated w/ brolucizumab 3mg & 45 CORE sub. w/ brolucizumab 6mg. These 107 sub. were treated in the extension w/ new formulation 6 mg brolucizumab. 43 subjects treated with aflibercept 2 mg in the CORE continued aflibercept.
Groups:
- Brolucizumab - Overall Extension Study: Subjects treated with brolucizumab 3 mg or brolucizumab 6 mg in the Core study. All subjects received IVT injection at the extension Baseline, Week 8 and, depending on disease activity as assessed by the investigator, at Week 16 or Week 20.
- Aflibercept: Subjects previously treated with aflibercept 2 mg in the Core study continued to receive aflibercept 2mg IVT injection at the extension Baseline, Week 8 and Week 16 to maintain the masking in the extension trial.
Period: Overall Study
Arm/Group | Brolucizumab - Overall Extension Study | Aflibercept
Started | 107 | 43
Completed (Completed exWeek 24) | 106 | 42
Not Completed | 1 | 1
Not completed — Death | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Extension safety set includes all subjects who entered the extension study and received at least one injection of study treatment in this extension study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brolucizumab - Overall Extension Study | Aflibercept | Total
Number analyzed (Participants) | 107 | 43 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.6 (8.63) | 77.9 (9.20) | 79.8 (8.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 22 | 91
  Male | 38 | 21 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 6 | 17
  Not Hispanic or Latino | 95 | 37 | 132
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Ocular and Non-Ocular Treatment Emergent Adverse Events
Description: Number of participants with ocular and non-ocular treatment emergent events with the new formulation brolucizumab 6 mg in this extension trial up to week 24 vs. the corresponding last 6 months of brolucizumab treatment in the Core trial >= 2%. Safety assessment of the new formulation brolucizumab 6 mg was based on a within-patient comparison with the last 6 months of corresponding Core safety data. Missing brolucizumab data were imputed using last observation carried forward (LOCF).
Time Frame: Up to Week 24
Population: Brolucizumab extension safety set included subjects who received at least one injection of brolucizumab 6mg. Data was presented descriptively for only brolucizumab in line with the study objective. No formal hypothesis testing was planned.
Measure: Number; unit: Participants
Groups:
- Brolucizumab Overall Last 6 Months From Core Study: AEs with a start date on or after the date of Core study Week 68 visit were counted
Arm/Group | Brolucizumab - Overall Extension Study | Brolucizumab Overall Last 6 Months From Core Study
Number analyzed (Participants) | 107 | 107
Participants
  Ocular AEs | 20 | 25
  Non-Ocular AEs | 51 | 50

2. Secondary Outcome: Change of Loss in BCVA of 15 Letters or More From Extension Baseline at Each Post-baseline Visit
Description: Best-corrected visual acuity for the study eye was tested at all study visits in a sitting position using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing protocol at an initial testing distance of 4 meters. Outcome measure was prespecified for brolucizumab arm only. Neither patient selection process nor expected sample sizes supported a valid comparison between aflibercept and brolucizumab. The aflibercept arm was included only to maintain the masking in the extension trial. Data presented descriptively for only brolucizumab in line with study objective. No formal hypothesis testing was planned. Missing brolucizumab data were imputed using last observation carried forward (LOCF).
Time Frame: Extension Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
Population: Extension Data Set included all subjects who entered extension study and received at least one injection of study treatment. Assessment of the efficacy and safety of brolucizumab 6 mg was based on a within-patient comparison with the last 6 months of corresponding core study efficacy data serving as the reference.
Measure: Number; unit: Number of Participants
Groups:
- Brolucizumab 6 mg - 3 mg in Core Study: Subjects treated with brolucizumab 3 mg in Core study and given new formulation 6 mg in Extension study. All subjects received IVT injection at the extension Baseline, Week 8 and, depending on disease activity as assessed by the investigator, at Week 16 or Week 20.
- Brolucizumab 6 mg - 6 mg in Core Study: Subjects treated with brolucizumab 6 mg in Core study and given new formulation 6 mg in Extension study. All subjects received IVT injection at the extension Baseline, Week 8 and, depending on disease activity as assessed by the investigator, at Week 16 or Week 20.
Arm/Group | Brolucizumab 6 mg - 3 mg in Core Study | Brolucizumab 6 mg - 6 mg in Core Study | Brolucizumab - Overall Extension Study
Number analyzed (Participants) | 62 | 45 | 107
Number of Participants
  exWeek 4 (>=15 letters loss) | 2 | 0 | 2
  exWeek 8 (>=15 letters loss) | 4 | 0 | 4
  exWeek 12 (>=15 letters loss) | 4 | 0 | 4
  exWeek 16 (>=15 letters loss) | 6 | 0 | 6
  exWeek 20 (>=15 letters loss) | 4 | 0 | 4
  exWeek 24 (>=15 letters loss) | 3 | 0 | 3

3. Secondary Outcome: Change in BCVA From Extension Baseline at Each Post-baseline Visit
Description: Best-corrected visual acuity for the study eye was tested at all study visits in a sitting position using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing protocol at an initial testing distance of 4 meters. Outcome measure was prespecified for brolucizumab arm only. Neither the patient selection process nor expected sample sizes supported a valid comparison between aflibercept and brolucizumab. The aflibercept arm was included only to maintain the masking in the extension trial. Data was presented descriptively for only brolucizumab in line with the study objective. No formal hypothesis testing was planned. Missing brolucizumab data were imputed using last observation carried forward (LOCF).
Time Frame: Extension baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
Population: Extension Data Set included all subjects who entered extension study and received at least one injection of study treatment. Assessment of the efficacy of brolucizumab 6 mg was based on a within-patient comparison with the last 6 months of corresponding core-study efficacy and safety data serving as the reference.
Measure: Mean (Standard Deviation); unit: Letter read
Arm/Group | Brolucizumab 6 mg - 3 mg in Core Study | Brolucizumab 6 mg - 6 mg in Core Study | Brolucizumab - Overall Extension Study
Number analyzed (Participants) | 62 | 45 | 107
Letter read
  exWeek 4 | -1.3 (6.26) | 0.5 (3.81) | -0.5 (5.42)
  exWeek 8 | -1.7 (6.90) | -0.4 (4.29) | -1.2 (5.96)
  exWeek 12 | -2.7 (7.73) | -0.3 (5.17) | -1.7 (6.84)
  exWeek 16 | -3.9 (8.42) | 0.8 (5.36) | -1.9 (7.63)
  exWeek 20 | -3.4 (7.66) | 0.5 (7.34) | -1.8 (7.75)
  exWeek 24 | -2.0 (8.17) | 0.3 (6.79) | -1.0 (7.67)

4. Secondary Outcome: Patients With Positive q12w Treatment Status at Week 20
Description: The estimate for the proportion of patients with a positive q12w treatment status at Week 24 was derived from Kaplan Meier time-to-event analyses for the event 'first q8w-need'. The outcome of the Kaplan-Meier analysis was estimated probability for maintaining on q12w up to the Disease Activity Assessment (DAA) at exWeek 20. Outcome measure was prespecified for brolucizumab arm only. Neither the patient selection process nor expected sample sizes supported a valid comparison between aflibercept and brolucizumab. The aflibercept arm was included only to maintain the masking in the extension trial. Data was presented descriptively for only brolucizumab in line with the study objective. No formal hypothesis testing was planned. Missing brolucizumab data were imputed using last observation carried forward (LOCF).
Time Frame: Week 20
Population: Extension Data Set included all subjects who entered extension study and received at least one injection of study treatment. Assessment of the efficacy and safety of brolucizumab 6 mg was based on a within-patient comparison with last 6 months of corresponding core-study efficacy data serving as reference.
Measure: Number; unit: Percentage of patients
Groups:
- Brolucizumab 6 mg- 6 mg in Core Study: Subjects treated with brolucizumab 6 mg in Core study and given new formulation 6 mg in Extension study. All subjects received IVT injection at the extension Baseline, Week 8 and, depending on disease activity as assessed by the investigator, at Week 16 or Week 20.
Arm/Group | Brolucizumab 6 mg - 3 mg in Core Study | Brolucizumab 6 mg- 6 mg in Core Study | Brolucizumab - Overall Extension Study
Number analyzed (Participants) | 62 | 45 | 107
Percentage of patients | 63.3 | 63.1 | 63.3

5. Secondary Outcome: Change in Central Sub-Field Thickness (CSFT) From Extension Baseline at Each Post-baseline Visit
Description: Measurement of the central subfield thickness of the retina was assessed using Optical Coherence Tomography (OCT) at each visit for the study eye. Outcome measure was prespecified for brolucizumab arm only. Neither the patient selection process nor expected sample sizes supported a valid comparison between aflibercept and brolucizumab. The aflibercept arm was included only to maintain the masking in the extension trial. Data was presented descriptively for only brolucizumab in line with the study objective. No formal hypothesis testing was planned. Missing brolucizumab data were imputed using last observation carried forward (LOCF).
Time Frame: Extension Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
Population: Extension Data Set included all subjects who entered extension study and received at least one injection of study treatment. Assessment of the efficacy and safety of brolucizumab 6 mg was based on a within-patient comparison with the last 6 months of corresponding core-study efficacy data serving as the reference.
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Brolucizumab 6 mg - 3 mg in Core Study | Brolucizumab 6 mg- 6 mg in Core Study | Brolucizumab - Overall Extension Study
Number analyzed (Participants) | 62 | 45 | 107
micrometer
  exWeek 4 | -19.2 (39.29) | -17.5 (40.76) | -18.5 (39.74)
  exWeek 8 | -6.3 (25.47) | -18.9 (31.74) | -11.6 (28.82)
  exWeek 12 | -17.9 (43.07) | -28.9 (48.80) | -22.5 (45.66)
  exWeek 16 | -7.8 (31.94) | -11.7 (39.83) | -9.4 (35.35)
  exWeek 20 | -10.1 (59.04) | -15.3 (46.20) | -12.3 (53.84)
  exWeek 24 | -19.8 (37.67) | -24.6 (42.10) | -21.8 (39.47)

6. Secondary Outcome: Percentage of Subjects With Positive Anti-drug Antibody (ADA) Status for Brolucuzumab 6 mg in Extension
Description: Positive integrated anti-drug antibodies (ADA) status is defined as induced ADA status with ADA negative at pre-dose and a post-dose titer value of greater than or equal to 30 at any time point or boosted ADA status with ADA positive at pre-dose and a post-dose titer value increase by more than 3-fold (1 dilution) at any time point. Outcome measure was prespecified for brolucizumab arm only. Neither the patient selection process nor expected sample sizes supported a valid comparison between aflibercept and brolucizumab. The aflibercept arm was included only to maintain the masking in the extension trial. Data was presented descriptively for only brolucizumab in line with the study objective. No formal hypothesis testing was planned. Missing brolucizumab data were imputed using last observation carried forward (LOCF).
Time Frame: Extension Baseline, Week 8, Week 16, Week 24
Population: Extension Data Set included all subjects who entered extension study and received at least one injection of study treatment. Assessment of efficacy and safety of brolucizumab 6 mg was based on a within-patient comparison with last 6 months of corresponding core-study efficacy data serving as the reference.
Measure: Number; unit: Percentage of participants
Arm/Group | Brolucizumab - Overall Extension Study
Number analyzed (Participants) | 107
Percentage of participants | 54

ADVERSE EVENTS:
Time Frame: From first treatment in the extension study, through study completion, to an average of 24 weeks. Adverse events and serious adverse events were collected for the maximum actual duration of treatment exposure and follow up for a participant per the protocol for approximately 6 months.
Description: Adverse events were recorded for AEs that started during the extension study, and AEs started during the Core study that were ongoing at ext. baseline. Safety assessment of broluizumab 6 mg was based on a within-patient comparison w/the last 6 months of corresponding Core safety data serving as reference. Adverse Events were obtained from subjects and observations by the Investigator as outlined in the study protocol. This analysis set includes all subjects who received at least 1 IVT injection.
Groups:
- Brolucizumab 6mg Overall Extension Study: Subjects treated with brolucizumab 3 mg or brolucizumab 6 mg in the Core study. All subjects received IVT injection at the extension Baseline, Week 8 and, depending on disease activity as assessed by the investigator, at Week 16 or Week 20.
- Brolucizumab Overall Last 6 Months Core Study: AEs with a start date on or after the date of Core study Week 68 visit were counted.
- Aflibercept 2 mg: Subjects previously treated with aflibercept 2 mg in the Core study continued to receive aflibercept 2mg IVT injection at the extension Baseline, Week 8 and Week 16 to maintain the masking in the extension trial.
Arm/Group | Brolucizumab 6mg Overall Extension Study | Brolucizumab Overall Last 6 Months Core Study | Aflibercept 2 mg
All-Cause Mortality (participants affected / at risk) | 1/107 | 0/107 | 0/43
Serious Adverse Events (participants affected / at risk) | 7/107 | 7/107 | 10/43
Other Adverse Events (participants affected / at risk) | 12/107 | 14/107 | 13/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6mg Overall Extension Study (N=107) | Brolucizumab Overall Last 6 Months Core Study (N=107) | Aflibercept 2 mg (N=43)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 1
Retinal artery occlusion - Study eye (Eye disorders) | 1 | 0 | 0
Retinal vein occlusion - Study eye (Eye disorders) | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6mg Overall Extension Study (N=107) | Brolucizumab Overall Last 6 Months Core Study (N=107) | Aflibercept 2 mg (N=43)
Cataract - Fellow eye (Eye disorders) | 1 | 1 | 3
Neovascular age-related macular degeneration - Fellow eye (Eye disorders) | 2 | 2 | 3
Nasopharyngitis (Infections and infestations) | 5 | 4 | 3
Urinary tract infection (Infections and infestations) | 4 | 6 | 6
Haematuria (Renal and urinary disorders) | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-09-27): https://cdn.clinicaltrials.gov/large-docs/74/NCT03386474/SAP_000.pdf
  • Study Protocol (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT03386474/Prot_001.pdf